CLINICAL TRIAL: NCT04329286
Title: Platelet Changes in Cases of Chronic Iron Over Load
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Jakleen Merzek Lowiz, principal investigator, Assiut University
Other Study IDs: Platelet changes
Record Dates: First submitted 2020-03-29; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Platelet Changes in Cases of Iron Overload

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Iron demand: The average daily demand to fit the cell biological metabolism is balanced between intake and lost which about 1-2 mg.

DETAILED DESCRIPTION:
Iron demand: The average daily demand to fit the cell biological metabolism is balanced between intake and lost which about 1-2 mg. One unit of packed red blood cells contains approximately 200-250 mg of iron.Thus, patients who arereceiving an average of 2 to 4 units of blood monthly willhave an iron intake of 5000to 10 000 mg of iron per year. Iron overload(IO) A condition in which the body takes up and stores more iron than it needs from any cause. Iron overload constitutes a major problem in patients receivingregular blood transfusion. Patients with β-thalassemia,sickle cell anemia, and congenital and refractory anemiasonchronic transfusion programs accumulate iron in variousbody organs. Untreated iron overload will eventually lead todamage of the liver, endocrine organs, and most seriously theheart(1).Acquired platelet function defect might be one of thecomplications of iron overload. This could occur indirectlythrough the effect of iron load on the liver and other organsor might occur due to effect of iron load on platelet functiondirectly. Dleteriouscomlications contributed by chemical reactive deregulated iron may affect cellular homeostasis systematically lead to tissue and organ damage when this toxicity occurred in blood cells ,alteration of peripheral hematological profile concerning erythrocyte,leucocyte and Platelet. On the other hand, acquired platelet function defects are classified broadly into defects that are intrinsic or extrinsic to the platelets. Acquired platelets defect are due to medications, medical conditions, underlying hematologic diseases, and are more frequent than inherited causes of platelets defects. (2) Platelet function is also influenced by changes in membranefluidity that has an important role in the expressionof platelet receptors and in modulating the activity ofproteins like phospholipase C or proteinkinase C(3). Ithas been shown (4) that changes in membrane fluidityare associated to altered aggregation/agglutination functionof freshly prepared platelets. The platelet aggregationresponse is modified by monovalent cations (whichalter fibrinogen binding) and monovalent anions thatenhance hydroxyl radicals production of platelets inducing platelet activation (5) Reactive oxygen species(ROS) are involved in integrin aIIbb3 activation(6,7). Moreover, bursts of ROS are generated in platelets exposed to thrombin (8). We herein report the case of a patient with acquired plateletfunction defect associated with iron overload as a consequenceof chronic blood transfusion. Therefore, we emphasizethe necessity of further studies to confirm directcorrelation between iron overload as a causative agent andplatelets dysfunction. And we recommend screening forplatelet function in patients receiving chronic blood transfusionaiming at possible prevention of any lifethreateningbleeding.

One of the most commonly used laboratorymarkers to early characterize platelet functionis the mean platelet volume (MPV). Increasedplatelet volume mayindicate its greater content ingranules, showing a platelet activation also betteraggregation and more reactive than the ordinarysize one. Limited study and the inconsistent resultare available regarding the platelet function studyin IO complicated condition. Higher MPV wasidentified in heterozygous beta-thalassemiapatientswith no correlation with cardiovascularrelatedrisks( 9). However, but in line with this study, adefect in platelet aggregation indicated by ahyporeactivityof platelet after induction withADP, ristocetin, and collagen was showed in majorthalassemia children patients

ELIGIBILITY:
Inclusion Criteria:

* Patients around age of 6 to 18 years
* Patients with thalassemia disease

Exclusion Criteria:

* - Patients less than 6 years and more than 18 years.

  * Patients with sever inflammatory disease.
  * Patients with any malignant disease.
  * Patients take steroid or bone marrow suppression drugs.
  * Patients with aplastic anemia or pancytopenia.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Platelet Changes in Cases of Iron Overload(IO)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Platelet Changes in Cases of Iron Overload(IO) | 1year
  Platelet Changes in Cases of Iron Overload(IO)

REFERENCES:
- [Background] Hoffbrand AV, Taher A, Cappellini MD. How I treat transfusional iron overload. Blood. 2012 Nov 1;120(18):3657-69. doi: 10.1182/blood-2012-05-370098. Epub 2012 Aug 23. PMID 22919029
- [Background] Vlasic N, Medow MS, Schwarz SM, Pritchard KA Jr, Stemerman MB. Lipid fluidity modulates platelet aggregation and agglutination in vitro. Life Sci. 1993;53(13):1053-60. doi: 10.1016/0024-3205(93)90258-5. PMID 8366768
- [Background] Wachowicz B, Olas B, Zbikowska HM, Buczynski A. Generation of reactive oxygen species in blood platelets. Platelets. 2002 May;13(3):175-82. doi: 10.1080/09533710022149395. PMID 12180500
- [Background] Cikrikcioglu MA, Celik K, Ekinci I, Nasifov M, Toprak AE, Cetin G, Genc S. Mean Platelet Volume in Heterozygous Beta Thalassaemia. Acta Haematol. 2017;137(2):100-105. doi: 10.1159/000455813. Epub 2017 Feb 17. PMID 28208125